CLINICAL TRIAL: NCT00005598
Title: A Phase II Trial of 5-Azacytidine (NSC #102816) and Ethyol (Amifostine) in the Treatment of Adults With Myelodysplastic Syndromes
Brief Title: Azacitidine Plus Amifostine in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067711; P30CA046592 (NIH); CCUM-9906 (Other: University of Michigan Cancer Center PRC); NCI-T99-0069
Record Dates: First submitted 2000-05-02; First posted 2003-12-16 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Myelodysplastic Syndromes
Keywords: refractory anemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory | interventions — Amifostine; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: azacitidine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Amifostine may improve blood counts in patients with myelodysplastic syndrome. Combining azacitidine with amifostine may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of azacitidine plus amifostine in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate to azacitidine plus amifostine in patients with myelodysplastic syndromes. II. Evaluate the toxicity of this treatment regimen in these patients. III. Assess the rate of progression to acute myeloid leukemia and overall survival in these patients treated with this regimen. IV. Evaluate the relationship between response status and cytogenetics, FAB class, ras mutations, and the presence of nonclonal hematopoiesis with this treatment regimen in these patients. V. Assess the effect of this treatment regimen on the number of bone marrow hematopoietic progenitor cells in these patients. VI. Evaluate neutrophil adhesion and chemotaxis in these patients before and after this treatment regimen.

OUTLINE: Patients receive amifostine IV over 1-3 minutes on days 8, 10, 12, 15, 17, 19, 22, 24, and 26 plus azacitidine subcutaneously on days 1-7. Treatment repeats every 28 days for 4 courses. Patients who achieve complete remission receive an additional 3 courses, and patients who achieve hematologic improvement or partial remission continue treatment until disease progression or unacceptable toxicity. Patients are followed until death.

PROJECTED ACCRUAL: A total of 17-32 patients will be accrued for this study within approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cytologically confirmed myelodysplastic syndrome (MDS) Intermediate 1, 2, or high risk disease OR Low risk disease with one of the following: Symptomatic anemia requiring transfusion for at least 3 months prior to study Symptomatic thrombocytopenia requiring platelet transfusion Platelet count less than 50,000/mm3 Absolute neutrophil count less than 1,000/mm3 with an infection Stable disease for 1 month with no progression to acute myeloid leukemia Declined or not eligible for allogeneic bone marrow transplant (alloBMT) No prior treatment of MDS with chemotherapy or alloBMT No prior leukemia or more than 30% myeloblasts in the bone marrow

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: 0-2 Life expectancy: Greater than 4 months Hematopoietic: See Disease Characteristics Hepatic: Bilirubin less than 1.5 times normal (unless due to hemolysis or ineffective erythropoiesis) AST and ALT less than 2 times normal Renal: Creatinine less than 1.5 times normal Cardiovascular: No uncontrolled or severe congestive heart failure Pulmonary: Serum CO2 greater than 18 mmHg Other: No uncorrected folate or vitamin B12 deficiency HIV negative No other medical or psychiatric illness that would preclude study At least 3 years since prior nonleukemic malignancy Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 1 month since prior interferon, interleukin-3, or interleukin-11 At least 1 month since prior epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF) No concurrent hematologic growth factors Chemotherapy: See Disease Characteristics Prior chemotherapy for nonleukemic malignancy allowed No prior azacitidine Endocrine therapy: At least 1 month since prior corticosteroids or danazol No concurrent steroids Radiotherapy: Prior radiotherapy for nonleukemic malignancy allowed Surgery: Not specified Other: No prior antithymocyte globulin or cyclosporine No prior amifostine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2001-12 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry P. Erba, MD, PhD, Study Chair — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States